CLINICAL TRIAL: NCT02085902
Title: Does the Use of Ropivacaine Facilitates Cholecystectomy by Laparoscopy in Ambulatory Surgery?
Acronym: VesiRop
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHD 079-13
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cholecystectomy; Laparoscopy
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard anesthesia (No Intervention)
- standard anesthesia with ropivacaine (Experimental): ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine
  Arms: standard anesthesia with ropivacaine

SUMMARY:
Since the recommendations of the French Society of Digestive Surgery 2010, cholecystectomy can be performed as outpatient surgery. This approach is difficult in many centers because of post operative pain and nausea/vomiting.

The use of postoperative morphine may be responsible for the state of nausea. The use of ropivacaine allows a reduction of the morphine consumption and thus may allow the patient to have their surgery as an outpatient.

Currently, ropivacaine is used randomly during the investigators surgeries. Initially, it was used for the infiltration holes trocar. In recent years, ropivacaine is used for the reduction of intra-abdominal postoperative pain. Its use is made of parietal surgery ( hernia ) in cholecystectomy and colonic surgery. This mode of administration is allowed to view the many publications made on this subject. Its use in the investigators daily surgery, however, has not been evaluated in ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* Programmed Cholecystectomy
* Laparoscopy
* Man and woman
* ≥ 18
* ASA 1 or 2
* Not living alone
* Patient receiving social security coverage
* Signature of Informed Consent Form

Exclusion Criteria:

* Cholecystectomy emergency
* Patient minor
* Pregnant woman (pregnancy test) or during breastfeeding
* Conversion to laparotomy
* Patient anticoagulant curative dose
* Living alone
* Patient addict
* Peptic Ulcer
* Refusal to enter the protocol
* Chronic requiring analgesics long-term
* Immunosuppression
* Long-term Treatment with corticosteroids
* Discovery intraoperative calculation in the bile duct
* Contraindication to ropivacaine (see cons-indications to ropivacaine)
* Hypersensitivity to study treatment or concomitant medications anesthesia
* Cardiac or unbalanced epileptic patients (due to the risk of cardiovascular and neurological local anesthetics)
* Patients ASA ≥ 3
* Patient <50 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time to discharge patient after surgery | 6 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Dr, Study Director — CHD Vendée La Roche sur Yon
Locations (1):
- Centre hospitalier départemental Vendée, La Roche-sur-Yon, France

REFERENCES:
- [Result] Abet E, Orion F, Denimal F, Brau-Weber AG, de Kerviler B, Jean MH, Boulanger G, Dimet J, Comy M. Interest of Using Ropivacaine for Outpatient Laparoscopic Cholecystectomy: Prospective Randomized Trial. World J Surg. 2017 Mar;41(3):687-692. doi: 10.1007/s00268-016-3797-2. PMID 27872974